CLINICAL TRIAL: NCT02386904
Title: Prospective, Interventional, Single Arm Study in Outpatients Undergoing Sigmoidoscopy for Evaluation of Efficacy and Safety of Kleen Enema 120ml (Phosphate Enema)
Brief Title: Safety and Therapeutic Efficacy of Phosphate Enema (Kleen Enema) in Patients Undergoing Sigmoidoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nabiqasim Industries (Pvt) Ltd (Industry)
Collaborators: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: • KLEE-EFF-002-01
Record Dates: First submitted 2015-03-07; First posted 2015-03-12 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phosphate Enema (Experimental): Phosphate Enema consisting on Monobasic Sodium Phosphate (USP) 19.2 gm /120 ml and Dibasic Sodium Phosphate (USP) 7.2 gm/120 ml Dosage Form: Enema Frequency: One time; 30 minutes before Sigmoidoscopy
  Interventions: Drug: Phosphate Enema (Kleen® Enema)

INTERVENTIONS:
Drug: Phosphate Enema (Kleen® Enema) — 120ml (single bottle) administered via rectal route before 30min of sigmoidoscopy .
  Other Names: Brand name is Kleen® Enema

SUMMARY:
The Purpose of the study is to determine the efficacy of Kleen Enema® (Phosphate Enema) for bowel preparation in out-patients under going sigmoidoscopy procedure and to evaluate the safety behavior of Kleen Enema® in outpatients requiring sigmoidoscopy

DETAILED DESCRIPTION:
Safety and therapeutic efficacy of Phosphate enema (Kleen Enema®) in patients undergoing sigmoidoscopy. Prospective, interventional, single arm study in patients undergoing day care sigmoidoscopy for evaluation of efficacy and safety of Kleen Enema®(120ml phosphate enema); manufactured by Nabiqasim Industries (Pvt) Ltd, Karachi, Pakistan.

Methods &Material:

Study will be conducted in patients undergoing sigmoidoscopy in day care at Dow University of Health Sciences, Ojha campus, Karachi. Each subject will receive the single dose of investigational drug (phosphate enema 120ml). Objectives of the study

* To determine the efficacy of Kleen Enema® for bowel preparation in out-patients undergoing to sigmoidoscopy procedure.
* To evaluate the Safety of Kleen Enema® in outpatients requiring sigmoidoscopy.

Rationale of the Study:

This would be helpful to determine the efficacy and safety of investigational product in local population.

Study Condition :

The study will be conducted in outpatients admitted for day care sigmoidoscopy requiring left sided bowel preparation for procedure. Each subject will receive the single dose of investigational drug (phosphate enema 120ml). Patient will remain in fasting condition at least 6 hours before procedure and half an hour after recovery from sedation; after this patient can take normal diet.

Ethical Considerations:

The study will be conducted after the approval by an Institutional review board of Dow University of Health Sciences, Karachi and in accordance to declaration of Helsinki, International Conference of Harmonization - Good Clinical Practices and Pakistan Good Clinical Practices guidelines to protect the rights and safety of human subjects as participants in the study.

Duration of study :

Study duration for primary efficacy end point evaluation will be the time period till sigmoidoscopy procedure is completed and patient is discharged from day care. While patient will come again for follow-up visit. Whole study will be completed in five months, after Institutional Review Board approval.

Sample Size:

Investigational drug will be administered to 40 Patients.The data of at least 35 patients will be included for efficacy study. While all enrolled patients who receive a single dose of study product will be included for safety evaluation.

Screening procedure Out patients visiting gastroenterology Out Patient Department requiring sigmoidoscopy will undergo screening procedure. Medical examination, history, vital signs, electrolytes test (Ca, Phosphate, Sodium and potassium levels) and CBC test will be performed. However the normal procedure and conditions required for sigmoidoscopy will be followed.

Drug administration Method for rectal enema:

Study patients should lay on left side with both knees bent, arms at rest.Remove protective shield from the enema container. With steady pressure, gently insert enema comfort tip into anus with nozzle pointing towards navel. Squeeze bottle until nearly all liquid is expelled. Discontinue use if resistance is encountered. Forcing the enema can result in injury.Return enema to carton for disposal. Generally, 2 to 5 minutes are sufficient to obtain the desired effect maximum to 30 minutes. Study subject may have an urge to evacuate the bowel.

Confinement :

After sigmoidoscopy is completed, patients will be monitored in the recovery room of endoscopy suite till patients are out of sedative effect.Safety Assessment Health assessment, including vital signs, physical examination and clinical laboratory testing (electrolyte test and CBC) will be performed at baseline; before sigmoidoscopy and electrolyte will be repeated within 10-30 minutes after dosing. Patients will be monitored after drug administration to determine any adverse events. Patients are encouraged to report any unusual feeling or adverse event to endoscopy research staff or research assistant. Patients will be monitored for pruritus, dehydration, nausea,vomiting, abdominal pain, abdominal distension, diarrhea, gastrointestinal pain and any other adverse

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female; aged 18-60 years.
2. Out-patients admitted for day care sigmoidoscopy requiring left sided bowel preparation
3. Able to understand the informed consent, answer the questions either independently or with someone helps

Exclusion Criteria:

1. In-patients undergoing sigmoidoscopy or as emergency procedures.
2. Immunosuppressed patients.
3. Patients with electrolyte imbalance or disturbance, Hyperphosphatemia, Hypocalcemia, Hypokalemia, Hypernatremia, Metabolic acidosis.
4. Patients having nausea, vomiting, diarrhea at the time of investigational drug administration.
5. Patients administering the medications known to affect renal perfusion, function, or hydration(Renal failure or acute kidney injury)
6. Patients taking diuretics or other medications within two days prior to the procedure which may alter electrolytes
7. Patients with known hypersensitivity to any ingredient of the study drug/phosphate.
8. Patients requiring colostomy.
9. Conditions causing decreased gastric motility, e.g.,Suspected intestinal obstruction,Paralytic ileus Anorectal stenosis, Imperforate anus, Congenital or acquired megacolon
10. Undiagnosed gastrointestinal pathology, e.g. Symptoms of appendicitis, intestinal perforation or active inflammatory bowel disease, Undiagnosed rectal bleeding, Dehydration and generally in all cases where absorption capacity is increased or elimination capacity is decreased
11. Patients with any neuropathy, renal impairment, liver diseases, diabetes mellitus, Hypertension and any Cardiovascular disease,History of asthma, glaucoma, or raised intraocular pressure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Excellent Preparation for Sigmoidoscopy (efficacy) | 30 minutes after administration of the Enema
  i. Small amounts of faecal material in scattered locations removable by suctioning and not preventing satisfactory visualisation of bowel mucosa; ii. Excellent preparation, no faecal material.

CONTACTS AND LOCATIONS:
Overall Officials: Hafeezullah Shaikh, FCPS, MBBS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- National Institute of Liver and GI diseases, DUHS, Karachi, Sindh, Pakistan